CLINICAL TRIAL: NCT02510170
Title: Fetal and Maternal Head Circumference During Pregnancy
Brief Title: Fetal and Maternal Head Circumference During Pregnancy in Israeli Population
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: COM150035CTIL
Record Dates: First submitted 2015-07-19; First posted 2015-07-29 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-01

CONDITIONS: Maternal-Fetal Relations; Microcephaly
Keywords: Fetus; Skull; ultrasonography
MeSH Terms: conditions — Microcephaly

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: no intervention

SUMMARY:
In this study, measurements of fetal and maternal head circumference will be collected. This data will be presented in table or graph form. The effect of maternal head circumference on fetal head circumference will be evaluated and presented in either formula or graph form.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Valid first trimester sonogram

Exclusion Criteria:

* Women under 18 years of age
* Women over 40 years of age
* Multi fetal pregnancy
* No accurate dating of pregnancy age
* Participant non compliance or cannot complete contact details
* Technical difficulty measuring fetal or maternal skull
* Abnormal fetal or maternal skull
* Familial hereditary disease, mental retardation
* Chronic maternal illness
* Maternal on chronic medication
* Abnormal screening test during current pregnancy
* Abnormal sugar metabolism or Hypertension during current pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fetal head circumference (millimeters) | 14 through 40 weeks pregnancy
  Israeli fetal population. Will be reported in table and / or graph form

SECONDARY OUTCOMES:
Relationship of fetal head circumference (mm) to maternal head circumference (mm) | 14 through 40 weeks pregnancy where applicable
  Calculating effect of maternal head circumference on fetal head circumference during pregnancy and adjusting (Formula) fetal head circumference normal values (+/- 2SD)
Maternal head circumference (millimeters) | age 18 through 40
  Israeli maternal population. Will be reported in table and / or graph form

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Health Center - Lev Tel-Aviv, Tel Aviv, Israel